CLINICAL TRIAL: NCT07039994
Title: Early Palliative Care in Patients With Advanced Lung Cancer Using an e-Health Ecosystem: a Randomized, Controlled, and Blinded Clinical Trial
Brief Title: Early Palliative Care in Patients With Advanced Lung Cancer Using an e-Health Ecosystem
Acronym: AIRPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jesús González (Other Government)
Collaborators: Institut Català d'Oncologia (Other); Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Sponsor-Investigator, Jesús González, MD, PhD, Instituto de Salud Carlos III
Organization: Instituto de Salud Carlos III (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AIRPAL-010521; PR274/21 (Other: Independent review board)
Record Dates: First submitted 2025-06-02; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Palliative Care; e-Health; Telemedicine; Early Treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Experimental group - e-Health follow-up, a combined system using ICT and in-person care. It includes spontaneous use (symptom tracking, messages, reminders via app) and scheduled use:
  * Good symptom control: Basic Telematic Evaluation (BTE) at 1 month. If stable, videoconference at 2 months, BTE at 3 months, and in-person visit at 4 months.
  * Poor symptom control: BTE at 1 week. If warning signs appear, a nurse evaluates by phone and may adjust treatment, schedule a visit (in-person or video), or refer to emergency care. In-person visit by need or after 1 month.
  Control group - Standard follow-up:
  * Good control: In-person visit every 4 weeks.
  * Poor control: Nurse calls at 1 week to assess and decide on treatment changes, visits, or referral. In-person visit by need or after 1 month.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-health follow-up (Experimental)
  Interventions: Other: E-health intervention
- Standard follow-up (Active Comparator)
  Interventions: Other: Standard intervention

INTERVENTIONS:
Other: Standard intervention — Routine intervention in the service:
  * Good control: In-person visit every 4 weeks.
  * Poor control: Nurse calls at 1 week to assess and decide on treatment changes, visits, or referral. In-person visit by need or after 1 month.
  Arms: Standard follow-up
Other: E-health intervention — Combined system using ICT and in-person care. It includes spontaneous use (symptom tracking, messages, reminders via app) and scheduled use:
  * Good symptom control: Basic Telematic Evaluation (BTE) at 1 month. If stable, videoconference at 2 months, BTE at 3 months, and in-person visit at 4 months.
  * Poor symptom control: BTE at 1 week. If warning signs appear, a nurse evaluates by phone and may adjust treatment, schedule a visit (in-person or video), or refer to emergency care. In-person visit by need or after 1 month.
  Arms: E-health follow-up

SUMMARY:
Palliative care has long been associated primarily with end-of-life support. However, its scope is much broader. As highlighted in the Hastings Center Report, the purposes of medicine include not only curing disease but also preventing illness, relieving suffering, caring for patients, avoiding preventable deaths, and ensuring a peaceful death when unavoidable. Palliative care plays a vital role in achieving all of these goals. In addition to pain and symptom management, it addresses the prevention of complicated grief, the emergence of severe symptoms (e.g., constipation, delirium), the inappropriate use of end-of-life treatments, and offers specialized care for incurable diseases.

This model of care follows a multidimensional and multidisciplinary approach, focusing on the person beyond the illness and addressing emotional, social, spiritual, and practical needs. Recent studies have shown that early integration of palliative care within routine oncology improves symptom control, emotional well-being, and coping with the illness. Furthermore, it enhances quality of life for both patients and their families, reduces healthcare resource usage, and does not increase overall health expenditure.

Such early integration also facilitates discussions about end-of-life issues, promotes advance care planning, and supports improved home-based palliative care. Additionally, it has been associated with fewer aggressive treatments and a positive impact on patient survival.

Systematic symptom assessment leads to earlier and more effective management. In this context, information and communication technologies (ICTs) have shown promise in enabling remote monitoring and care delivery. These tools can enhance quality of life, improve treatment adherence, reduce emergency visits, and positively influence survival. However, existing studies have limitations, such as small sample sizes and lack of evaluator blinding.

The COVID-19 pandemic emphasized the need for physical distancing and accelerated the development of remote healthcare systems. Some specialized cancer centers, like the Institut Català d'Oncologia, have implemented functional multidisciplinary units for each cancer type. These units consist of various specialists (medical oncologists, radiation oncologists, surgeons, radiologists, pathologists, advanced practice nurses, palliative care professionals, etc.) who collaboratively decide the best course of treatment. A key role within these units is the reference nurse, assigned to each patient, who acts as a main point of contact, available for in-person or phone consultations.

One major improvement in recent years has been the integration of palliative care clinics within oncology departments. Best practices now emphasize early palliative intervention based on patient complexity and needs. While no universal definition exists, most studies define "early palliative care" as involvement by a palliative team within the first three months following a diagnosis of advanced cancer. This approach is supported by multiple scientific societies. Nevertheless, challenges such as limited resources, accessibility barriers, and increasing in-person demand near the end of life remain significant obstacles.

Among advanced cancers, lung cancer stands out due to its high prevalence and poor prognosis. It is characterized by frequent and unpredictable symptoms, requiring flexible and responsive follow-up. Adapting care to patients' changing needs could improve quality of life, optimize resources, and reduce the frequency of in-person visits.

This study proposes the integration of early palliative care with an e-Health ecosystem, reflecting the global push to bring care into the homes of vulnerable patients using modern technology. Evidence for the impact of ICTs in palliative care remains limited, and existing studies are generally of low quality. To date, only one registered trial (NCT03375489) has explored e-Health in early palliative care. Unlike that study, this research offers a scalable model tailored to patient complexity, alongside a comprehensive cost-utility evaluation (e.g., fewer in-person visits, emergency care use, and patient transfers to care centers).

This is the first international clinical trial of its kind in palliative care. It is a multicenter, randomized, controlled trial with blinded third-party evaluation. The hypothesis is that an e-Health ecosystem with ICT tools will improve access, early detection, monitoring, and remote palliative intervention for lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced NSCLC (stage III or IV) with criteria for early palliative intervention*, seen in the initial palliative care consultation.
* Patients or primary caregivers with internet proficiency and access to computer and telephone equipment.
* Patients with ECOG performance status 0-3

  * For the purposes of this study, patients with the following conditions will be considered candidates for early palliative care: a tumor diagnosis ≤3 months prior to diagnosis and one or more of the following criteria: average pain poorly controlled with opioids (VAS score ≥4); dyspnea on minor exertion; patients <60 years of age; emotional distress (HADS ≥10); family fragility; functional limitation (Barthel <60); history or use of drugs; and the presence of ethical or existential dilemmas (Llorens et al., 2017; Tuca et al., 2019).

Exclusion Criteria:

* Patients who do not meet criteria for early palliative intervention.
* Patients with severe cognitive impairment or psychiatric impairment that prevents proper evaluation.
* Patients who do not speak or understand Catalan or Spanish adequately.
* Patients who, at the first visit, are in a serious clinical condition that prevents proper evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2028-03-24 (Estimated); Study Completion 2028-07-24 (Estimated)

PRIMARY OUTCOMES:
FACT-L | Baseline, 3, 6, 9 and 12 months
  Functional Assessment of Cancer Therapy-Lung Minimum and maximum values: 0-136 worst to best quality of life

SECONDARY OUTCOMES:
ESAS-r | Baseline, 3, 6, 9 and 12 months
  Edmonton Symptom Assessment System Minimum and maximum values: 0-1, meaning no symptom to 11 symptoms scored 0-10 /110
HADS | Baseline, 3, 6, 9 and 12 months
  Hospital Anxiety and Depression Scale Ranges from 0-42. Higher scores indicate greater anxiety and/or depression symptoms.
EQ-5D-3L | Baseline, 3, 6, 9 and 12 months
  European Quality of Life Scale Scale Ranges from 5-15, with 5 being best Quality of Life
ARMS | Baseline, 3, 6 ,9 and 12 months
  Adherence to Refills and Medications Values ranges from 12 to 48, being 12 maximum adherence to refills
CTCAE | Baseline, 3, 6, 9 and 12 months
  Common Toxicology Criteria for Adverse Events Grade 1. Mild: Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2. Moderate: Minimal, local, or noninvasive intervention indicated; limitation of age-appropriate instrumental Activities of Daily Living (ADLs).
  Grade 3. Severe or medically significant but not immediately life-threatening: Hospitalization or prolongation of hospitalization indicated; disabling; limits self-care ADLs.
  Grade 4. Life-threatening consequences: Urgent intervention indicated. Grade 5. Death related to adverse event (AE).
Opioid dose | Baseline, 3, 6, 9 and 12 months
  Daily oral morphine equivalent dose, in miligrams/day
Hospitalization rate | 3, 6, 9 and 12 months
PSCRCM | Baseline, 3, 6, 9 and 12 months
  Patient Satisfaction with Cancer-Related Care Measure Scale between 18 to 90, being 18 maximum satisfaction
Charlson Index | Baseline, 3, 6, 9 and 12 months
  Comorbidity Scale ranging between 0 to 32, being 0 no comorbidities and 32 all comorbidities of the test
PPS | Baseline, 3, 6, 9 and 12 months
  Palliative Performance Scale Percentage (100-10), being 100 normal functionality and 10 patient completely bedridden, no possibility of work, complete depence for selfcare, only able to ingest solids and sleepy or in a coma
ECOG | Baseline, 3, 6, 9 and 12 months
  Eastern Cooperative Oncology Group (functionality) Grade 0: The patient is completely asymptomatic and is able to perform normal work and daily life activities.
  Grade 1: The patient has symptoms that prevent them from doing strenuous work but is able to carry out normal daily activities and light work. The patient only stays in bed during nighttime sleep hours.
  Grade 2: The patient is unable to perform any work and has symptoms that force them to stay in bed for several hours during the day, in addition to nighttime, but not exceeding 50% of the day. The individual manages most of their personal needs independently.
  Grade 3: The patient needs to be bedridden for more than half of the day due to symptoms. They require assistance with most activities of daily living, such as dressing.
  Grade 4: The patient needs to be bedridden 100% of the day and requires help with all activities of daily living, such as personal hygiene, moving in bed, and even feeding.
  Grade 5: Patient deceased.
Pfeiffer questionaire | Baseline, 3, 6, 9 and 12 months
  Cognitive State Scale between -1 to 9, being -1 intact and 9 severe impairment
BPI | Baseline, 3, 6, 9 and 12 months
  Brief Pain Inventory Scale between 0 to 10 to determine maximum, minimum and mean pain in the last 24 hours, being 0 no pain and 10 maximum pain Percentage to determine interference of pain with activities, or to determine pain improvement after medication
Age | Baseline registry
  Number
Sex | Baseline
  Male or female
Type of cancer | Baseline
  Adenocarcinoma, scamous carcinoma or indiferentiated
Stage | Baseline
  IA, IB, IIA, IIB, IIIA, IIB, IIIC, IVA or IVB
Aim of the onco-specific treatment | Baseline
  Curative, palliative, non-decided or non onco-specific treatment
Type of onco-specific treatment | Baseline, 3, 6, 9 and 12 months
  Chemotherapy, radiotherapy, surgery, Inmunotherapy, Targeted Therapy or non-onco-specific treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jesús González Barboteo, MD, PhD, Principal Investigator — Catalan Institute of Oncology (ICO)
Locations (2):
- Spain (2):
  - Catalan Institute of Oncology, Badalona, Barcelona
  - Catalan Institute of Oncology, L'Hospitalet de Llobregat, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided